CLINICAL TRIAL: NCT06817330
Title: the Effect of a MUsic Intervention on poStictal Agitation in Electroconvulsive Therapy Patients: the MUSE Trial
Brief Title: The Effect of a Music Intervention on Postictal Agitation in Electroconvulsive Therapy Patients
Acronym: MUSE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Erasmus Medical Center (Other)
Collaborators: Parnassia Groep (Other)
Responsible Party: Principal Investigator, Markus Klimek, Vice-Charmain Department of Anesthesiology, Director Residency Training Program Department of Anesthesiology, Erasmus Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NL86074.078.24
Record Dates: First submitted 2025-01-29; First posted 2025-02-10 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-12

CONDITIONS: Music Intervention; Electroconvulsive Therapy Treated Patients; Agitation on Recovery From Sedation
Keywords: music; postictal agitation; electroconvulsive therapy
MeSH Terms: interventions — Control Groups

STUDY DESIGN:
Intervention Model Description: Multi-center prospective randomized controlled trial with a parallel design.
Masking Description: Due to the nature of the study and the music intervention, it is not possible to blind participants and investigators.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group, listening to recorded music (Experimental): Recorded music, with headphones, for 30 minutes directly before ECT and 12 minutes directly after ECT.
  Interventions: Other: Intervention group, listening to recorded music
- Control group, headphones with no music (Other): Headphones with no music or sound, for 30 minutes directly before ECT and 12 minutes directly after ECT.
  Interventions: Other: Control group, headphones with no music

INTERVENTIONS:
Other: Intervention group, listening to recorded music — Participants in the group receiving music will be offered a tablet with several pre-created playlists. When the patient has made a selection, they will listen to music via headphones for 30 minutes before each ECT treatment session. The headphones will be removed and the music stopped after the 30 minutes. After active ECT treatment, the headphones will be put back on the patient and the music played for another 12 minutes while the patient is recovering and moved to the recovery room. If patients protest against the music and/or headphones, the researcher will ask them to put the headphones back on. If the patient still protests after asking to put the headphones back on, this will be written down by the researcher, with the amount of time without the (control) intervention noted. No coercion will be used during the whole study process.
  Arms: Intervention group, listening to recorded music
Other: Control group, headphones with no music — The control group will wear headphones without music for the same duration as the music group (30 minutes before ECT and 12 minutes after ECT) to reduce bias and achieve a similar level of background-noise dampening.
  Arms: Control group, headphones with no music

SUMMARY:
This study will investigate the effect of music on postictal agitation when played peri-interventionally for patients undergoing electroconvulsive therapy for severe depression.

DETAILED DESCRIPTION:
Postictal agitation (PIA) is a fairly common adverse effect after electroconvulsive therapy (ECT) treatment that, when present, predicts other complications such as retrograde amnesia. Multiple studies have suggested that a music intervention in the context of surgery significantly reduces pre-operative anxiety, as well as the need for sedatives and analgesic medication. Pretreatment anxiety is common for ECT patients and is a known predictor of PIA. Currently, there is no preventative treatment for PIA. Given the beneficial effects of music demonstrated in similar hospital settings combined with its easy implementation and lack of side effects, the investigators hypothesize that music listening can lower the incidence and severity of PIA among patients undergoing ECT therapy, thereby also reducing post-treatment cognitive impairment. Therefore, the objective of the study is to assess the effect of music on postictal agitation when played peri-interventionally for patients undergoing electroconvulsive therapy for severe depression.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing ECT treatment for depression (including depression as part of bipolar disorder)
* Adult patients (≥18 years)
* Hypnotic agent used is etomidate
* Sufficient understanding of the Dutch language (in judgement of the attending physician or researcher)
* Written informed consent by patient or legal representative

Exclusion Criteria:

* Significant impaired hearing (defined as unable to communicate verbally or listen to music)
* Severe neurological condition (defined as interfering with the ability to process music)
* Patients receiving ECT for treatment of schizophrenic disorders

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 92 (Estimated)
Dates: Start 2025-11-25 (Actual); Primary Completion 2027-02-28 (Estimated); Study Completion 2027-02-28 (Estimated)

PRIMARY OUTCOMES:
Presence or absence of postictal agitation | First 30 minutes post-ECT session
  The primary outcome measure is the presence or absence of postictal agitation (PIA). All patients will be screened for PIA using the RASS (Richmond Agitation-Sedation Scale), a 10-point scale, indicating alertness and responsiveness, taking less than 20 seconds to perform. The scale ranges from -5 (deep sedation) to +4 (extreme agitation), with positive scores indicating agitation (higher score is more agitation so worse outcome) relevant for diagnosing PIA. Screening for PIA will be conducted after the first six ECT treatments by a nurse or medical student who will monitor the patient for 30 minutes in the recovery room. PIA is defined as agitation leading to a score of +1 or greater on the RASS during this period. Patients scoring less than +1 will be recorded as having no PIA for that session. Nurses and medical students will receive training on using the RASS scale, documented in the training log and side delegation file.

SECONDARY OUTCOMES:
Severity of postictal agitation | First 30 minutes post-ECT session
  All patients will be screened for PIA using the RASS (Richmond Agitation-Sedation Scale), a 10-point scale, indicating alertness and responsiveness, taking less than 20 seconds to perform. The scale ranges from -5 (deep sedation) to +4 (extreme agitation), with positive scores indicating agitation (higher score is more agitation so worse outcome) relevant for diagnosing PIA. Patients will screen positive for PIA if the RASS is at least +1. Mild PIA is characterized by a RASS score of +1, while moderate and severe PIA are indicated by scores of ≥ +2. A RASS score of at least +2 is associated with a greater risk of danger to the patient and/or staff.
Duration of postictal agitation | First 30 minutes post-ECT session
  All patients will be screened for PIA using the RASS (Richmond Agitation-Sedation Scale), a 10-point scale, indicating alertness and responsiveness, taking less than 20 seconds to perform. The scale ranges from -5 (deep sedation) to +4 (extreme agitation), with positive scores indicating agitation (higher score is more agitation so worse outcome) relevant for diagnosing PIA. The duration of PIA will be measured as the time from the highest observed RASS score to a RASS score of zero. A longer duration is longer agitation so a worse outcome. PIA duration is a predictor of retrograde amnesia following ECT, with shorter durations being desirable.
Pretreatment anxiety | Directly before and after the 30-minute music or control intervention prior to ECT session
  Patients will be screened for pretreatment anxiety using the VAS-A, a validated self-rating measurement ranging from 0 (not at all anxious) to 10 (extremely anxious).
Music listening behavior | Directly before the 30-minute music or control intervention prior to the ECT session
  Before each intervention/ECT session, patients will be asked if and how long they listened to music the day before treatment.
Duration of recovery | Directly after ECT-session, till leaving recovery room and/or medically ready to be discharged, up to 2 hours post-ECT session
  Recovery duration will be measured as the total time spent in the recovery room after ECT. The time that the patient is deemed medically ready to be discharged (but has not yet left) will also be noted.
Peri-treatment medication requirement | From 24 hours prior to ECT session until leaving the recovery room, up to 2 hours post-ECT session
  Peri-treatment medication requirement includes all medication used from 24 hours before ECT until leaving the recovery room, with dosage corrected for body weight (mg/kg) for medications such as antipsychotics, benzodiazepines, mood stabilizers, and opioids.
Cognitive impairment | Within 7 days prior to ECT course and 2 and 90 days after completing ECT course
  Cognitive impairment will be assessed using the MoCA (Montreal Cognitive Assessment), a scale ranging from 0-30. Lower scores mean more cognitive impairment, so worse outocmes. Anything below 26 is a sign of cognitive impairment. The MoCA will be administered within 7 days before the first ECT treatment (baseline) and during follow-up at 2 and 90 days after the patient's completion of the full ECT course.
Severity of depression | Within 7 days prior to ECT course and weekly during the ECT course (up to 4 months)
  Depression severity will be measured before the start of the ECT course and weekly during the course using the HDRS (Hamilton Depression Rating Scale, range 0-52) or the MADRS (Montgomery-Åsberg Depression Rating Scale, range 0-60). For both scales, higher ratings mean more depression so a worse outcome. To avoid overburdening the severly depressed patients in this study with additional questionnaires, both scales will be used in accordance with standard care procedures at the participating centers. The HDRS and MADRS scales are correlated and can be converted between each other, which will be done during the analysis phase of the study.

CONTACTS AND LOCATIONS:
Overall Officials: Markus Klimek, MD, PhD, Principal Investigator — Erasmus Medical Center
Locations (2):
- Netherlands (2):
  - Erasmus Medical Center, Rotterdam
  - Antes Parnassia Group, Rotterdam

IPD SHARING:
Plan to Share IPD: No
Data will only be shared upon request. This decision will be made by the principal investigator.

REFERENCES:
- [Background] Leucht S, Fennema H, Engel RR, Kaspers-Janssen M, Szegedi A. Translating the HAM-D into the MADRS and vice versa with equipercentile linking. J Affect Disord. 2018 Jan 15;226:326-331. doi: 10.1016/j.jad.2017.09.042. Epub 2017 Sep 27. PMID 29031182
- [Background] Graff V, Wingfield P, Adams D, Rabinowitz T. An Investigation of Patient Preferences for Music Played Before Electroconvulsive Therapy. J ECT. 2016 Sep;32(3):192-6. doi: 10.1097/YCT.0000000000000315. PMID 27075143
- [Background] Schuur G, Verdijk JPAJ, Ten Doesschate F, van Wingen GA, van Waarde JA. Severe Postictal Confusion After Electroconvulsive Therapy: A Retrospective Study. J ECT. 2023 Mar 1;39(1):34-41. doi: 10.1097/YCT.0000000000000866. Epub 2022 May 25. PMID 36825989
- [Background] Andrade C, Arumugham SS, Thirthalli J. Adverse Effects of Electroconvulsive Therapy. Psychiatr Clin North Am. 2016 Sep;39(3):513-30. doi: 10.1016/j.psc.2016.04.004. Epub 2016 Jun 25. PMID 27514303
- [Background] Ertman M, van der Valk Bouman ES, Clephas PRD, Birkenhager TK, Klimek M. Prognostic Factors and Incidence for Postictal Agitation After Electroconvulsive Therapy: A Systematic Review and Meta-analysis. J ECT. 2025 Mar 1;41(1):17-26. doi: 10.1097/YCT.0000000000001032. Epub 2024 Aug 22. PMID 39105589
- [Derived] van der Valk Bouman ES, Ertman M, Koopmans MR, van der Vlugt-Molenaar JJB, Heijnen WTCJ, van Groen JC, Korstanje JW, Birkenhager TK, Klimek M. Effect of peri-interventional music on postictal agitation in electroconvulsive therapy patients (MUSE): protocol for an open-label multicentre randomised controlled trial in the Netherlands. BMJ Open. 2025 Dec 10;15(12):e105979. doi: 10.1136/bmjopen-2025-105979. PMID 41371746